CLINICAL TRIAL: NCT02330094
Title: Gabapentin for Headache in Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William D. Freeman, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-005288
Record Dates: First submitted 2014-12-24; First posted 2015-01-01 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aSAH; SAH
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin capsules 100 mg ter in die (TID), 200 mg TID, 300 mg TID, 400 mg TID, 600 mg TID, 900 mg TID.
  Interventions: Drug: Gabapentin
- Control (Placebo Comparator): Placebo capsules 100 mg ter in die (TID), 200 mg TID, 300 mg TID, 400 mg TID, 600 mg TID, 900 mg TID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin capsules will be administered orally and titrated from 100 mg - 900 mg TID based on the patient's numeric pain score and creatinine clearance.
  Both groups will receive other standard of care pain medications.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — Placebo capsules will be administered orally and titrated from 100 mg - 900 mg TID based on the patient's numeric pain score and creatinine clearance.
  Both groups will receive other standard of care pain medications.
  Arms: Control

SUMMARY:
The purpose of this study is to see how much gabapentin will reduce headaches associated with subarachnoid hemorrhage (SAH) and to reduce the amount of narcotic pain medication prescribed.

DETAILED DESCRIPTION:
The investigators plan to use gabapentin (GBP), an FDA approved non-narcotic pain medication for neuropathic pain, which is also an alpha-2-delta (A2DR) receptor analogue to reduce the pain and decrease the need for narcotics in patients with aneurysmal subarachnoid hemorrhage (aSAH). GBP has been shown to decrease neuropathic and non-neuropathic pain in a variety of perioperative and postoperative conditions. A2DR affinity also has some neuroprotective effect in animal data. The investigators plan to conduct a prospective, double-blinded, randomized trial to further assess GBP-associated reductions in narcotic use and pain scores compared to the non-GBP (placebo) arm. To accomplish this aim, the investigators plan to randomize 20 aSAH patients with headache to either GBP and standard of care pain treatment versus placebo and standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Have aneurysmal subarachnoid hemorrhage (aSAH) diagnosed by CT scan of the brain and/or angiogram evidence of intracranial aneurysm (CTA or digital subtraction angiogram or MRA)
3. Have symptomatic headache
4. Able to swallow and verbalize pain score
5. No known allergy to gabapentin or fentanyl
6. Numeric pain score ≥ 5
7. Ability to provide written personal consent

Exclusion Criteria:

1. Gabapentin use prior to SAH admission
2. Renal failure with creatinine clearance less than 30 mL/min
3. Unable to receive standard of care pain medications
4. Pregnant or breastfeeding patients
5. History of severe depression defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Freeman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Dhakal LP, Turnbull MT, Jackson DA, Edwards E, Hodge DO, Thottempudi N, Kamireddi P, Akinduro OO, Miller DA, Meschia JF, Freeman WD. Safety, Tolerability, and Efficacy of Pain Reduction by Gabapentin for Acute Headache and Meningismus After Aneurysmal Subarachnoid Hemorrhage: A Pilot Study. Front Neurol. 2020 Jul 28;11:744. doi: 10.3389/fneur.2020.00744. eCollection 2020. PMID 32849209
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Gabapentin capsules 100 mg ter in die (TID), 200 mg TID, 300 mg TID, 400 mg TID, 600 mg TID, 900 mg TID.
  Gabapentin: Gabapentin capsules will be administered orally and titrated from 100 mg - 900 mg TID based on the patient's numeric pain score and creatinine clearance.
  Both groups will receive other standard of care pain medications.
- Control: Placebo capsules 100 mg ter in die (TID), 200 mg TID, 300 mg TID, 400 mg TID, 600 mg TID, 900 mg TID.
  Placebo: Placebo capsules will be administered orally and titrated from 100 mg - 900 mg TID based on the patient's numeric pain score and creatinine clearance.
  Both groups will receive other standard of care pain medications.
Period: Overall Study
Arm/Group | Gabapentin | Control
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gabapentin: Gabapentin capsules 100 mg TID, 200 mg TID, 300 mg TID, 400 mg TID, 600 mg TID, 900 mg TID.
  Gabapentin: Gabapentin capsules will be administered orally and titrated from 100 mg - 900 mg TID based on the patient's numeric pain score and creatinine clearance.
  Both groups will receive other standard of care pain medications.
- Control: Placebo capsules 100 mg TID, 200 mg TID, 300 mg TID, 400 mg TID, 600 mg TID, 900 mg TID.
  Placebo: Placebo capsules will be administered orally and titrated from 100 mg - 900 mg TID based on the patient's numeric pain score and creatinine clearance.
  Both groups will receive other standard of care pain medications.
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Control | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (10.2) | 49.8 (11.6) | 51.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16
Chronic Pain [Count of Participants; unit: Participants] — Chronic pain is ongoing pain that lasts for more than 6 months.
  Participants | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Average Numeric Pain Score
Description: Pain was measured on a Visual Analogue Scale (VAS) rated from 0-10, where 0 was no pain and 10 was the worst pain imaginable. The numeric pain score was measured every 4 hours and the total score over 24 hours was averaged as the daily numeric pain score. The daily scores were then averaged over a 7 day period for a single average pain score.
Time Frame: baseline through day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 8 | 8
score on a scale | 5.2 (1.9) | 5.8 (1.5)
Statistical Analysis 1: Comparison: Gabapentin vs Control; Test type: Superiority; p = 0.7, t-test, 2 sided

2. Primary Outcome: Average Narcotic Consumption
Description: The amount of narcotics administered, averaged over a 7 day period, calculated in total morphine equivalents (ME).
Time Frame: baseline through day 7
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 8 | 8
milligrams | 19.4 (14.8) | 20.2 (13.1)
Statistical Analysis 1: Comparison: Gabapentin vs Control; Test type: Superiority; p = 0.79, ANOVA

3. Secondary Outcome: Pain Control Satisfaction Questionnaire
Description: The Brigham and Women's Hospital Management of Post-operative Pain Patients discharge questionnaire (BWQ) was used to measure pain control satisfaction. The questionnaire was modified and transformed into a uniform scale so all numbers were on the same direction. Subjects were asked to answer six questions on a score of 0-5, for a total possible range of 0-30. A lower score indicated a better outcome (less pain) and higher pain control satisfaction and a higher score indicated a worse outcome (more pain) and lower pain control satisfaction.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 8 | 8
score on a scale | 14 (4.1) | 12.6 (2.9)
Statistical Analysis 1: Comparison: Gabapentin vs Control; Test type: Superiority; p = 0.66, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of time the subject was in the Neuro Intensive Care Unit, which was an average of 7 to 14 days.
Arm/Group | Gabapentin | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=8) | Control (N=8)
Nausea (General disorders) | 1 (1) | 1 (1)
Agitation (General disorders) | 1 (1) | 1 (1)
Delirium (General disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT02330094/Prot_SAP_000.pdf